CLINICAL TRIAL: NCT00165048
Title: Selective COX-II Inhibitor as a Palliative Therapy in Patients With R1 or R2 Resection for Disseminated Stomach Cancer - A Multi-Centre Prospective Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2001.462-T
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-09

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — rofecoxib

INTERVENTIONS:
Drug: Vioxx (Rofecoxib)

SUMMARY:
The purpose of this study is to investigate the effect of selective COX-II inhibitor in patients with regionally disseminated stomach cancer treated by palliative resection (so called R1 or R2 gastrectomy).

DETAILED DESCRIPTION:
Cyclo-oxygenase (COX) is a family of enzymes regulating the conversion of arachidonic acid to prostaglandins. COX-II is an inducible enzyme, which expresses excessively when there are stimuli such as inflammation or hypergastrinaemia. Up to 40% of patients with stomach cancer are found to have disseminated disease during surgical exploration. While palliative resection could offer a marginal benefit in the survival of these patients, almost all patients will die of progression of disease within a short time span. Palliative chemotherapy has been used in the past. However, there is no evidence that the chemotherapy can confer any survival advantages, and the side-effects and toxicity of the treatment may indeed compromise the quality of life of these patients. With a better understanding of the relation between COX-II and stomach cancer, it may be possible to suppress the progression of the residual cancer cells after the palliative resection by giving the patients selective COX-II inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Stomach cancer with peritoneal or lymphatic spread beyond the scope of curative resection
* Palliative resection can be performed
* Normal RFT

Exclusion Criteria:

* Solid organ metastases
* Poor performance status
* On long-term aspirin or NSAID
* Renal or hepatic dysfunction
* Bleeding disorder
* Hypersensitive to COX-II inhibitors/aspirin/NSAID
* No history of myocardial infarct or stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206
Dates: Start 2004-10

PRIMARY OUTCOMES:
Symptom-free susrvival and the quality of life score within the two years of study period.

SECONDARY OUTCOMES:
Overall survival in long-term.

CONTACTS AND LOCATIONS:
Overall Officials: Enders K.W. Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Combined Gastro-intestinal Cancer Clinic, Hong Kong, China